CLINICAL TRIAL: NCT05004402
Title: Pelvic Floor Muscle Function, Pelvic Floor Dysfunction and Diastasis Recti Abdominis in Postpartum Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PN/56/2021
Record Dates: First submitted 2021-07-22; First posted 2021-08-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pelvic Floor Disorders; Diastasis Recti
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primiparous women: Primiparous women after vaginal delivery

SUMMARY:
Background: Pregnancy and childbirth are factors that affect a woman's pelvic floor. Pelvic floor disorders (PFD) often occur in the perinatal period. Symptoms and difficulties related to urinary continence and/or pelvic organ prolapse significantly affect daily activities, including physical activity, but also the quality of life and sexual activity. Patient education that includes both the anatomy and function of the pelvic floor, as well as information on the prevention of PFD during pregnancy and postpartum is an important part of the prevention of these dysfunctions. Diastasis recti abdominis (DRA) is another common musculoskeletal issue related to pregnancy and postpartum period. In addition to the cosmetic consequences, it can be associated with abdominal pain, the occurrence of pelvic floor dysfunction and a negative correlation with the image of a woman's own body.

Material and Methods: Primiparous women after vaginal delivery will be invited to this study. The study will consist of three stages. First phase (baseline measurements) will take place at the hospital and the following assessments will be performed: pelvic floor muscle palpation examination (PERFECT scheme, OXFORD scale, Reissing scale), palpation and ultrasound examination of diastasis recti abdominis. After 12-16 weeks postpartum participants will complete questionnaires about pelvic floor dysfunctions and diastasis recti and their impact on quality of life. Third part, 12-16 weeks postpartum, the pelvic floor muscle examination, palpation and ultrasound examination of diastasis recti abdominis will be repeated.

Objectives: The aim of this study is to assess the function of the pelvic floor muscles, prevalence of pelvic floor dysfunctions and diastasis recti abdominis in the primiparous women postpartum. Our secondary objective will be investigation if there are any prognostics factors during the early postpartum period, that can indicate higher risk of PFD and/or DRA 3 months postpartum.

Expected results: Results of this study will inform about prevalence of pelvic floor dysfunctions and diastasis recti in primiparous women in Poland. Additionally, we hope to obtain predictors suggesting pelvic floor or abdominal muscles dysfunction 3 months postpartum. Prevention of pelvic floor disorders may contribute to the early identification of problems and reduce cost of treatment of unrecognized dysfunction. To our knowledge this will be the first study in this area conducted in Poland.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery between 38-42 weeks of pregnancy
* First delivery
* Agreement to participate
* Good command of spoken and written Polish

Exclusion Criteria:

* Contraindications for the examination of the pelvic floor muscles (postpartum hematoma of the perineum, extensive perineal swelling, perineal wound dehiscence, bladder catheterization).
* Lack of consent to participate in the study
* Lack of good command of spoken and written Polish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primiparous women after vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Palpation examination of pelvic floor muscles with the use of PERFECT Scheme | 24-72 hours postpartum
  Assesment of pelvic floor muscles with the use of PERFECT Scheme.
Palpation examination of pelvic floor muscles with the use of PERFECT Scheme | 12-16 weeks postpartum
  Assesment of pelvic floor muscles with the use of PERFECT Scheme.
Ultrasound measurement of inter-recti distance (IRD) | 24-72 hours postpartum
  Measurement of inter-recti distance (IRD) using the ultrasound.
Ultrasound measurement of inter-recti distance (IRD) | 12-16 weeks postpartum
  Measurement of inter-recti distance (IRD) using the ultrasound.
Polish version of the Pelvic Floor Distress Inventory (PFDI-20) | 12-16 weeks postpartum
  Condition-specific questionnaire will be used to assess how pelvic floor disorders affect quality of life. It consist of 3 scales, 20 questions. Every scale is scored from 0- no distress to 100 - the greatest distress. The scores from 3 scales are summarized to achieve summary score (0-300).
Polish version of the Pelvic Floor Impact Questionnaire short form 7 (PFIQ-7) | 12-16 weeks postpartum
  Condition-specific questionnaire, will be used to assess impact of pelvic floor disorders on quality of life (daily activities, relationships and emotions). It consists of 3 scales which are scored 0-100. The results from 3 scales are summarized to achieve the summary score (0-300). Higher numbers indicate greater impact.
Polish Version of the Female Sexual Function Index (FSFI) | 12-16 weeks postpartum
  Assessment of sexual function in women, in 6 domains (desire, arousal, lubrication, orgasm, satisfaction, pain) scored 0-6. The summarized maximum score is 36. Results ≤27,50 indicate risk for sexual dysfunction.

SECONDARY OUTCOMES:
Palpation evaluation of pelvic muscle tone with Reissing scale | 24-72 hours postpartum
  Assessment of muscle tone. Reissing scale for palpation evaluation of muscle tone with use of 7-level grade where -3 means hypotonic, 0 -normotonus and +3 hypertonic muscles.
Palpation evaluation of pelvic muscle tone with Reissing scale | 12-16 weeks postpartum
  Assessment of muscle tone. Reissing scale for palpation evaluation of muscle tone with use of 7-level grade where -3 means hypotonic, 0 -normotonus and +3 hypertonic muscles.
Palpable measurement of inter-recti distance (IRD) | 24-72 hours postpartum
  Palpable measurement of inter-recti distance (IRD) using electronic digital caliper.
Palpable measurement of inter-recti distance (IRD) | 12-16 weeks postpartum
  Palpable measurement of inter-recti distance (IRD) using electronic digital caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Starzec-Proserpio, PhD, Principal Investigator — Department of Midwifery, Centre of Postgraduate Medical Education, Warsaw, Poland
Locations (1):
- St. Sophia's Specialist Hospital, Warsaw, Poland